CLINICAL TRIAL: NCT06331000
Title: DIATRIM : Effect of One Year Elexacaftor-tezacaftor-ivacaftor Treatment on Glucose Tolerance Abnormalities in Adult Patients With Cystic Fibrosis.
Brief Title: Effect of One Year Elexacaftor-tezacaftor-ivacaftor Treatment
Acronym: DIATRIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9248
Record Dates: First submitted 2024-02-23; First posted 2024-03-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Elexacaftor-Tezacaftor-Ivacaftor; Glucose tolerance abnormalities
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with cystic fibrosis
  Interventions: Drug: elexacaftor-tezacaftor-ivacaftor treatment

INTERVENTIONS:
Drug: elexacaftor-tezacaftor-ivacaftor treatment — Effect of one year elexacaftor-tezacaftor-ivacaftor treatment on glucose tolerance abnormalities in adult patients with cystic fibrosis

SUMMARY:
The development of CFTR (cystic fibrosis conductance transmembrane regulator) modulators for people with cystic fibrosis (pwCF) and eligible for these treatments is a true therapeutic revolution. The major beneficial effect of CFTR modulators (CFTRm) on pulmonary function and the reduction of pulmonary exacerbations should have a considerable impact on the quality of life and patient's life expectancy. Data on the impact of CFTRm on glucose tolerance abnormalities are still very fragmentary. The investigators can think that their use, earlier and earlier in the history of the disease, will transform the evolutionary trajectories of patients on the respiratory, nutritional and metabolic levels.

Diabetes represents a major challenge in the management of pwCF because it is a factor in morbidity and mortality at all stages of the disease, from children to patients with terminal respiratory failure requiring lung transplantation. Early abnormalities in glucose tolerance observed in childhood, before the stage of diabetes, are also associated with poor pulmonary and nutritional outcomes. Experimental data suggest a positive effect of CFTRm on insulin secretion. However, investigators do not currently know the impact of CFTRm in patients with very early glucose disorders or at the stage of diabetes treated with insulin. Recently continuous glucose measurement (CGM) devices represent very effective tools for assessing abnormalities in glucose tolerance before the stage of diabetes and for monitoring patients treated with insulin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis aged over 18
* Patients treated for 1 year by elexacaftortezacaftor-ivacaftor
* Normal tolerant or intolerant to glucose or presenting with cystic fibrosis related diabetes treated or not with insulin
* Patient who had a continuous glucose monitoring in the 6 months before and 6 months after one year of treatment with elexacaftor-tezacaftor-ivacaftor

Exclusion Criteria:

* Patient not eligible for triple CFTR modulator
* Patient intolerant to triple corrector
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cystic fibrosis aged over 18, followed in cystic fibrosis ambulatory care services of 18 french centers
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Evaluate time in range of blood glucose variation >140 mg/dl during 2 weeks in a cohort of adult patients treated for one year with elexacaftor-tezacaftor-ivacaftor | time in range of blood glucose variation >140 mg/dl one year before and one year after the begining of elexacaftor-tezacaftor-ivacaftor treatment

SECONDARY OUTCOMES:
Evaluate other CGM parameters : time in range of blood glucose >180mg/dl ; >140mg/dl ; <70mg/dl ; 70-180 mg/dl ; 70-140mg/dl | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment
Marker of metabolic status: HbA1c (mmol/l) | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment
Marker of metabolic status: HbA1c (%) | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment
Marker of metabolic status: C-Peptid (µg/L) | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment
Marker of metabolic status: C-Peptid (nmol/L) | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment
Markers of nutritional status: Evaluation of weight monitoring (kg) | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment
Markers of nutritional status: Body Mass Index (BMI) | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment
Diabetes treatment (assess insulin needs) : mean glucose value per day (mg/dl) | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment
Assessment of respiratory function parameters : number of IV antibiotics | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment
Number patients with severe hypoglycaemia and serious adverse events | One year before and one year after the start of elexacaftor-tezacaftor-ivacaftor treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No